CLINICAL TRIAL: NCT04314973
Title: PaDAWAn: Parkinson's Disease - Adaptive Walking Assistance
Acronym: PaDAWAn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PaDAWAn
Record Dates: First submitted 2020-03-11; First posted 2020-03-19 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease
Keywords: Exoskeleton; Active Pelvis Orthosis
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evaluation sessions (Active Comparator): Patients will be evaluated while walking without wearing the robotic device, once before the intervention phase, once right after, and once a month after.
  Interventions: Other: Walking exercises
- Intervention phase (Experimental): Patients will walk with the robotic device, for 12 sessions of 10 min.
  Interventions: Device: Active Pelvis Orthosis

INTERVENTIONS:
Device: Active Pelvis Orthosis — Walking with the robotic device providing the assistive protocol.
  Arms: Intervention phase
Other: Walking exercises — Walking exercises without wearing the robotic device.
  Arms: Evaluation sessions

SUMMARY:
The goal of this study is to develop and validate a haptic assistive method in order to support walking in patients with Parkinson's disease, delivered to the patient's hips through a wearable robotic pelvis orthosis.

DETAILED DESCRIPTION:
None of the existing robotic devices used for gait rehabilitation in Parkinson's disease is wearable. Thanks to the wearable robotic pelvis orthosis we will use, the rehabilitation sessions can take place in an ecological environment.

The other advantage of the proposed assistance protocol is its adaptability: patients will feel their hips pattern to be "smoothed" by the robot, but they will keep the freedom of continuously steering their main movement variables (like stride frequency, duration, and length). A key measured metric will precisely rely on this variability between stride durations. Indeed, the degree of stride-to-stride variability was shown to reflect the patient's physiological state, and to be correlated with the stage of the disease.

Experimental trials will be conducted to assess both the assistive (i.e. the therapy effect during the therapy itself) and rehabilitative (i.e. effect after the therapy) natures of our protocol. The second main objective of this project will be the analysis of the effects of our protocol regarding the stride-to-stride variability of patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease diagnosis positive according to UK Brain Bank criteria
* Hoehn and Yahr score of 1 to 3
* Mini-mental state (MMSE) higher than 24
* Optimal drug treatment for at least 4 weeks at the time of inclusion
* No contraindication to physical exercising (ACSM criteria)

Exclusion Criteria:

* Not being able to understand French well enough
* Not being in the targeted age range

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Long-Range Autocorrelation (LRA) | From day 0 up to 8 weeks
  Assesses the variability between stride durations

SECONDARY OUTCOMES:
Unified Parkinson's disease rating scales (UPDRS) | From day 0 up to 8 weeks
  Assesses the disease stage and severity
Activities-Specific Balance Confidence Scale (ABC) | From day 0 up to 8 weeks
  Self reported measure of balance confidence in performing various activities
Balance Evaluation Systems Test (BESTest) | From day 0 up to 8 weeks
  The balance of subjects is tested during 6 postural control contexts
Gait analysis | From day 0 up to 8 weeks
  Average stride length and duration, gait symmetry, hips range of motion
Joint torques | From day 0 up to 8 weeks
  In order to assess the mechanical efforts associated to walking
Physiological Cost Index | From day 0 up to 8 weeks
  In order to assess the metabolic efforts associated to walking
System Usability Scale (SUS) | After 4 weeks
  Self reported measure of the fatigue and stress felt by patients

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otlet V, Vandamme C, Warlop T, Crevecoeur F, Ronsse R. Effects of overground gait training assisted by a wearable exoskeleton in patients with Parkinson's disease. J Neuroeng Rehabil. 2023 Nov 16;20(1):156. doi: 10.1186/s12984-023-01280-y. PMID 37974229